CLINICAL TRIAL: NCT01471730
Title: The ZEroPLASmaTrial (ZEPLAST): a Randomized, Controlled Trial on Transfusion Avoidance in High Transfusion-risk Cardiac Surgery Patients
Brief Title: The ZEro PLASma Trial (ZEPLAST): Avoidance of Fresh Frozen Plasma in Cardiac Surgery
Acronym: ZEPLAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Marco Ranucci, Director of Clinical Research in the Department of the Anesthesia and Intensive care, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7-020-MR; 2011-005223-40 (EudraCT Number)
Record Dates: First submitted 2011-11-07; First posted 2011-11-16 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Heart Disease
Keywords: Transfusions; Fresh Frozen Plasma; Fibrinogen; Prothrombin complex
MeSH Terms: conditions — Heart Diseases | interventions — Fibrinogen; Saline Solution; prothrombin complex concentrates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Saline solution (Placebo Comparator)
  Interventions: Drug: Saline solution
- Fibrinogen (Active Comparator)
  Interventions: Drug: Fibrinogen
- Prothrombin complex (Active Comparator)
  Interventions: Drug: Prothrombin complex

INTERVENTIONS:
Drug: Fibrinogen — All the patients randomized and not withdrawn will be tested 20 minutes before removal of aortic cross clamping with a Thromboelastometric fibrinogen test FIBTEM (Rotem) . They will all receive either human fibrinogen concentrate (according to the formula: (22 [mm] - MCF [mm]) * body weight [kg] / 140 [m] = whole g fibrinogen to be dosed as HFC) (treatment group) or placebo (control group). Study drug or placebo has to be administered after protamine.
  Other Names: RIASTAP
  Arms: Fibrinogen
Drug: Saline solution — Normal saline will be administered to control patients.
  Other Names: Placebo
  Arms: Saline solution
Drug: Prothrombin complex — After 15min from study drug administration and in presence of ongoing microvascular bleeding, we run a CT EXTEM. In case of prolonged CT time at EXTEM as long as 80 seconds [M1] , they will receive coagulation factors concentrates (Confidex) at a weight-based dose of 7 U/kg b.w. (treatment group) or placebo.
  Other Names: CONFIDEX
  Arms: Prothrombin complex

SUMMARY:
Prospective, randomized, double blind trial. The rationale of the study is the concept that fresh frozen plasma (FFP) is still largely used in cardiac surgery, despite the fact that prothrombin complexes and fibrinogen are available.The experimental hypothesis is that cardiac surgery patients may be operated with no use of FFP and with a coagulation factors replacement based on fibrinogen and prothrombin complexes (when needed).

Primary endpoint: Transfusion avoidance Secondary endpoints: Transfusion limitation, massive blood transfusion, bleeding.

Study population: high-risk adult cardiac surgery patients Sample size : 2 groups of 60 patients each

DETAILED DESCRIPTION:
Study design Randomized, placebo-controlled, double-blinded study Endpoints Primary: Transfusion avoidance of every allogeneic blood product Secondary: Reduction in the number of allogeneic blood products used, reduction in massive blood transfusion events incidence, reduction in postoperative bleeding.

Patient population This study is focused on the role of coagulation factors substitutes in avoiding transfusions. Therefore, the patient population should be composed by patients being at high-risk for transfusions due to bleeding and not to hemodilution. Moreover, bleeding should be primarily due to a coagulation factors deficiency, rather than to other causes (namely, drug-induced platelet dysfunction).

The major determinant of coagulation factors consumption during cardiac operations is the length of CPB. Only patients undergoing operations with a predictable CPB duration > 90 minutes will be admitted. This includes patients undergoing complex cardiac operations (double valve; CABG+valve; ascending aorta; adult congenital patients). Adult congenital patient may be of particular interest, since they usually have a preoperative reduced hepatic coagulation factors synthesis, due to venous stasis and polycythemia.

To avoid the effects of hemodilution in determining transfusional needs, patients with an expected lowest HCT < 23% during CPB will not be admitted to the study. This means excluding patients with a preoperative HCT < 35%, and patients with a small BSA (< 1.7 m2). Hemodilution during CPB will be checked, and in case of a HCT value < 23% the patient will be withdrawn from the study.

Power analysis and sample size

Data from our Institutional database (about 15,000 patients) have been retrieved according to the above reported selection criteria. 1,535 patients (10%) fulfill the randomization and no-withdrawal criteria.

Within this group, we could calculate the following outcome variables:

Variable Incidence Mean with SD Transfusion rate (any kind) 61% Packed red cells 57% FFP 31% Platelets 8% Big bleeders (> 800 mL) 20% Postoperative bleeding 560±501 Surgical revision 5.7%

Based on these data, we could perform a power analysis based on an alpha value of 0.05 and a beta value of 0.20. According to these values, the required number of patients to be enrolled varies according to the experimental hypothesis:

Transfusion rate control group Hypothesis for transfusion rate in treatment group Number of patients per each group Total number of patients 60% 30% 40 80 60% 35% 58 116 60% 40% 94 188

The study size will be 116 patients (58 per group).

Study protocol

Patients in the control group will receive the standard treatment available in our Hospital for blood management and hemostasis and coagulation control. This includes antifibrinolytic administration (tranexamic acid 15 mg/kg before CPB and 15 mg/kg after protamine) Patients in both groups will be transfused according to our standard protocol (attachment 1)

Randomization: sealed envelopes. Enveloped placed in the pharmacy. Preparation of the drug vs. placebo by a dedicated biologist. Blinded vials sent to the OR.

Dosing protocol

All the patients randomized and not withdrawn will be tested 20 minutes before removal of aortic cross clamping with a thromboelastometry fibrinogen test FIBTEM (Rotem) . They will all receive either human fibrinogen concentrate (according to the formula: (22 [mm] - MCF [mm]) * body weight [kg] / 140 [m] = whole g fibrinogen to be dosed as HFC) (treatment group) or placebo (control group). Study drug or placebo has to be administered after protamine.

After 15min from study drug administration and in presence of ongoing microvascular bleeding, we run a CT EXTEM. In case of prolonged CT time at EXTEM as long as 80 seconds [M1] , they will receive coagulation factors concentrates (Confidex) at a weight-based dose of 7 U/kg b.w. (treatment group) or placebo.

In presence of ongoing microvascular bleeding intraoperatively or during the first 6 hours in the ICU, the patients will be treated with other drugs and products to control bleeding according to our standard protocol (see "Transfusion protocol").

After dosing, a blood sample will be withdrawn, centrifuge, and frozen plasma will be stored for subsequent Thrombin Generation Test.

Blinding:

An unblinded biologist will follow the drug randomization process, open the sealed envelope, drug preparation, and ROTEM analysis.

All the other Investigators will be blinded.

Transfusion protocol

1. Definition of bleeding: Intraoperatively: delayed sterna closure due to microvascular bleeding Postoperatively: 2 mL/kg for 2 consecutive hours; or 1.5 ml/kg for 4 consecutive hours

Packed red cells will be transfused (one unit at a time) under the following conditions:

1. Always if Hb < 7 g/dL
2. Possible if Hb between 7 and 8 g/dL
3. Possible but with medical justification (hemodynamic instability; high oxygen extraction rate; signs of organ ischemia…) if Hb between 8 and 9 g/dL
4. Never if Hb ≥ 9 g/dL

Fresh frozen plasma in case of bleeding if

1. INR > 1.5
2. R time at TEG (with heparinase) > 12 minutes

Platelets in case of bleeding if

1. Platelet count < 50.000/mmc
2. Pre-treatment with thienopyridinies (not applicable in this study)

In case of intractable bleeding determining hemodynamic instability, and for all life-saving conditions, the above mentioned conditions may be not considered, and an empirical rescue therapy is allowed.

Funding This study will be funded internally with the IRCCS Policlinico San Donato Research Fund.

The drugs (fibrinogen concentrate and PCC) will be provided free of charge by CSL Behring, as well as the reagents for ROTEM analysis,

ELIGIBILITY:
Inclusion Criteria:

* The patients will be screened according to a modified TRUST1 Transfusion Score. This score attributes 1 point to each of the following conditions:

  * Hb level < 13.5 g/dL
  * Weight < 77 kg
  * Female sex
  * Age > 65 years
  * Non elective surgery
  * Serum creatinine > 1.36 mg/dL
  * Redo operation
  * Non isolated surgery
  * Factors are hemodilution-related factors, and will not be included. Non isolated surgery is mandatory for inclusion. Patients will be included in presence of at least 1 within the remaining 4 risk factors:
  * Age > 65 years
  * Non elective surgery
  * Serum creatinine > 1.36 mg/dL '8Redo operation INCLUSION CRITERIA (patients randomized)

    1. Combined cardiac operation with expected CPB duration > 90 minutes
    2. At least one additional risk factor within the following: Age > 65 years; Non elective surgery; Serum creatinine > 1.36 mg/dL; Redo operation

Exclusion Criteria:

1. Age < 18 years
2. Patients under thienopyridines
3. Known coagulopathy
4. Known autoimmune disorders
5. Participation in another RCT
6. Pregnancy
7. Emergency operation
8. Baseline HCT < 35%
9. Baseline Antithrombin < 80%
10. BSA < 1.7 m2

WITHDRAWAL CRITERION:

1. Lowest HCT on CPB < 23%
2. Transfusions during CPB

   * Patients randomized and not withdrawn will be DOSED with the investigational drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Avoidance of allogeneic blood products transfusion | 30 days
  Includes avoidance of packed red cells, FFP, platelet concentrates, cryoprecipitates

SECONDARY OUTCOMES:
Reduction in allogeneic blood products transfusions | 30 days
Massive blood transfusion | First postoperative 24 hours
  Number of patients experiencing blood transfusion of 7 RBC units or more in the first postoperative 24 hours.
Bleeding | First postoperative 12 hours
  Amount of postoperative bleeding that the patients experience in the first postoperative 12 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranucci, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, MI, Italy

REFERENCES:
- [Background] Rahe-Meyer N, Pichlmaier M, Haverich A, Solomon C, Winterhalter M, Piepenbrock S, Tanaka KA. Bleeding management with fibrinogen concentrate targeting a high-normal plasma fibrinogen level: a pilot study. Br J Anaesth. 2009 Jun;102(6):785-92. doi: 10.1093/bja/aep089. Epub 2009 May 2. PMID 19411671
- [Background] Solomon C, Pichlmaier U, Schoechl H, Hagl C, Raymondos K, Scheinichen D, Koppert W, Rahe-Meyer N. Recovery of fibrinogen after administration of fibrinogen concentrate to patients with severe bleeding after cardiopulmonary bypass surgery. Br J Anaesth. 2010 May;104(5):555-62. doi: 10.1093/bja/aeq058. Epub 2010 Mar 26. PMID 20348140
- [Background] Stanworth SJ, Brunskill SJ, Hyde CJ, McClelland DB, Murphy MF. Is fresh frozen plasma clinically effective? A systematic review of randomized controlled trials. Br J Haematol. 2004 Jul;126(1):139-52. doi: 10.1111/j.1365-2141.2004.04973.x. PMID 15198745
- [Background] Alghamdi AA, Davis A, Brister S, Corey P, Logan A. Development and validation of Transfusion Risk Understanding Scoring Tool (TRUST) to stratify cardiac surgery patients according to their blood transfusion needs. Transfusion. 2006 Jul;46(7):1120-9. doi: 10.1111/j.1537-2995.2006.00860.x. PMID 16836558
- [Background] Rahe-Meyer N, Solomon C, Winterhalter M, Piepenbrock S, Tanaka K, Haverich A, Pichlmaier M. Thromboelastometry-guided administration of fibrinogen concentrate for the treatment of excessive intraoperative bleeding in thoracoabdominal aortic aneurysm surgery. J Thorac Cardiovasc Surg. 2009 Sep;138(3):694-702. doi: 10.1016/j.jtcvs.2008.11.065. Epub 2009 May 17. PMID 19698858
- [Background] Bolliger D, Szlam F, Molinaro RJ, Rahe-Meyer N, Levy JH, Tanaka KA. Finding the optimal concentration range for fibrinogen replacement after severe haemodilution: an in vitro model. Br J Anaesth. 2009 Jun;102(6):793-9. doi: 10.1093/bja/aep098. Epub 2009 May 6. PMID 19420005
- [Derived] Ranucci M, Baryshnikova E, Crapelli GB, Rahe-Meyer N, Menicanti L, Frigiola A; Surgical Clinical Outcome REsearch (SCORE) Group. Randomized, double-blinded, placebo-controlled trial of fibrinogen concentrate supplementation after complex cardiac surgery. J Am Heart Assoc. 2015 Jun 2;4(6):e002066. doi: 10.1161/JAHA.115.002066. PMID 26037084